CLINICAL TRIAL: NCT03019666
Title: A Phase I Trial Testing NAM Expanded Haploidentical or Mismatched Related Donor Natural Killer (NK) Cells Followed by a Short Course of IL-2 for the Treatment of Relapsed/Refractory Multiple Myeloma and Relapsed/Refractory CD20+ Non-Hodgkin Lymphoma
Brief Title: Ph I Trial of NAM NK Cells and IL-2 for Adult Pts With MM and NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS057; MT2015-46 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Mantle-Cell Lymphoma; Follicular Lymphoma; Indolent B Cell Lymphoma; Primary Mediastinal Lymphoma; Lymphoplasmacytic Lymphoma
Keywords: MM; NHL; NK Cell; NK Cells
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multiple Myeloma (Experimental): After a lymphodepleting preparative regimen of cyclophosphamide and fludarabine, patients receive expanded NAM-NK cells followed by a short course of interleukin-2 (IL-2) to facilitate natural killer cell survival and expansion in vivo. Monoclonal antibodies and elotuzumab for Multiple Myeloma patients, will be administered prior to and after the natural killer cell infusion(s) to facilitate tumor targeting and antibody dependent cellular cytotoxicity (ADCC).
  Interventions: Biological: Nicotinamide Expanded Haploidentical or Mismatched Related Donor Natural Killer Cells
- Non-Hodgkin Lymphoma (Experimental): After a lymphodepleting preparative regimen of cyclophosphamide and fludarabine, patients receive expanded NAM-NK cells followed by a short course of interleukin-2 (IL-2) to facilitate natural killer cell survival and expansion in vivo. Monoclonal antibodies and rituximab for Non-Hodgkin Lymphoma patients, will be administered prior to and after the natural killer cell infusion(s) to facilitate tumor targeting and antibody dependent cellular cytotoxicity (ADCC).
  Interventions: Biological: Nicotinamide Expanded Haploidentical or Mismatched Related Donor Natural Killer Cells

INTERVENTIONS:
Biological: Nicotinamide Expanded Haploidentical or Mismatched Related Donor Natural Killer Cells — * Cyclophosphamide 40 mg/kg x 1 day on Day -5
  * Fludarabine 25 mg/m^2 x 3 days (Day -5, Day -4, day-3)
  Other Names: NAM-NK

SUMMARY:
This is a phase I trial with pilot expansion of HLA-haploidentical or HLA-mismatched related donor nicotinamide expanded-natural killer (NAM-NK) cell based therapy for patients with relapsed or refractory multiple myeloma (MM) or relapsed/refractory CD20-positive non-Hodgkin lymphoma (NHL). The primary endpoint of the study is to determine the maximum tolerated dose (MTD) of NAM-NK cells while maintaining safety.

ELIGIBILITY:
Patient Inclusion Criteria:

* ≥18 to ≤70 years of age
* Meets one of the following disease criteria:

  * Multiple Myeloma (MM) meeting one of the following:

    * relapsed/refractory disease after two lines of therapies, including a proteasome inhibitor (bortezomib, carfilzomib or ixazomib) and an immunomodulatory drug (thalidomide, lenalidomide or pomalidomide)
    * relapsed disease between 2-18 months of 1st autologous stem cell transplantation,
    * relapsed disease at least 4 months after allogeneic stem cell transplantation with no evidence of active graft versus host disease and no availability of donor lymphocyte infusion
    * measurable disease defined as serum IgG, A, M M-protein ≥ 0.5g/dL or serum IgD M-protein ≥ 0.5 g/dL, or urine M-protein ≥ 200 mg/24 hours
    * at least 4 weeks since plasmapheresis
    * at least 3 days between last corticosteroids and study treatment start
  * CD20-positive B-cell Non-Hodgkin Lymphoma (NHL)

    * CD20 expression confirmed by flow cytometry or immunohistochemistry and meeting one or more of the following:

      * evidence of relapsed/refractory disease that has failed conventional therapy and failed/not eligible/refused studies of a higher priority,
      * relapsed disease at least 60 days after autologous stem cell transplantation
      * relapsed disease at least 4 months after allogeneic stem cell transplantation with no evidence of active graft versus host disease and no availability of donor lymphocyte infusion
      * has measurable disease >1.5 cm in diameter
* HLA-haploidentical or mismatched related donor (aged 12 to 70 years) with donor/recipient match based on a minimum of intermediate resolution DNA based Class I typing of the A and B locus (at least 2/4 class I allele) and absence of recipient anti HLA antibodies against selected donor
* Karnofsky Performance Status ≥ 60% - appendix III
* Adequate organ function within 14 days of study registration (30 days for pulmonary and cardiac assessments) defined as:

  * Bone Marrow: Total white blood cell (WBC) count ≥ 3000/μL, absolute neutrophil count (ANC) ≥ 1000/μL, platelet count ≥ 75,000/μL and hemoglobin ≥ 8.0 g/dL - may be waived if abnormalities are due to disease related bone marrow involvement
  * Renal: creatinine ≤ 1.5 mg/dL or creatinine clearance ≥40mL/min using Cockcroft-Gault formula
  * Hepatic: ALT or AST ≤ 3 x upper limit of institutional normal (ULN), total bilirubin ≤ 1.5 x ULN
  * Pulmonary Function: oxygen saturation ≥ 90% on room air. If symptomatic or prior known impairment, pulmonary function ≥ 50% corrected DLCO and FEV1 is required
  * Cardiac Function: LVEF ≥ 40%, no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Calcium (MM only): Corrected calcium < 11.5 mg/dL within 2 weeks prior to enrollment
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to NAM-NK cell infusion (excluding preparative regimen pre-medications)
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
* Must have recovered from acute effects of prior therapy - at least 2 weeks should have elapsed since the last dose of chemotherapy
* Voluntary written consent

Patient Exclusion Criteria:

* Active, untreated CNS involvement
* Chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), or high-grade lymphomas (Burkittt's lymphoma/Lymphoblastic lymphoma)
* Pregnant or breastfeeding - The agents used in this study include those that fall under Pregnancy Category D - have known teratogenic potential. For elotuzumab arm: Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 14 days of study treatment start (24 hours prior to the start of elotuzumab)
* Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds)
* Class II or greater New York Heart Association Functional Classification criteria (appendix III) or serious cardiac arrhythmias likely to increase the risk of cardiac complications of cytokine therapy (e.g. ventricular tachycardia, frequent ventricular ectopy, or supraventricular tachyarrhythmia requiring chronic therapy)
* Active autoimmune disease requiring immunosuppressive therapy
* History of severe asthma, presently on chronic medications (a history of mild asthma requiring inhaled steroids only is eligible)
* New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Active uncontrolled bacterial, fungal, or viral infections - all prior infections must have resolved following optimal therapy
* Known hypersensitivity to any of the study agents used
* For MM patients only:

  * Prior radiotherapy within 2 weeks prior to the administration of study drug"
  * Surgery within 4 weeks
  * Chemo within 3 weeks (6 weeks for melphalan, or monoclonal antibodies)
* Received investigational drugs within the 14 days before 1st dose of study drug
* High titer of donor specific anti-HLA antibodies (MFI >1000)

DONOR INCLUSION CRITERIA:

* HLA-haploidentical or mismatched related donor/recipient match based on a minimum of intermediate resolution DNA based Class I typing of the A and B locus (at least 2/4 class I allele) and absence of recipient anti HLA antibodies
* 12 to 70 years of age - Priority should be given to age (<35 years), followed by HLA matching (haploidentical and if not available then fully mismatched donor).
* At least 40 kilogram body weight
* In general good health as determined by the evaluating medical provider
* Adequate organ function defined as:

  * Hematologic: hemoglobin, WBC, platelet within 10% of upper and lower limit of normal range of test (gender based for hemoglobin),
  * Hepatic: ALT < 2 x upper limit of normal,
  * Renal: serum creatinine < 1.8 mg/dl
* Performance of a donor infectious disease screen panel including CMV Antibody, Hepatitis B Surface Antigen, Hepatitis B Core Antibody, Hepatitis C Antibody, HIV PCR, HIV ½ Antibody, HTLVA ½ Antibody, Rapid Plasma (RPR) Treponema , Trypanosoma Cruzi (T. Cruzi), HCV by NAT, HIV by NAT and WNV (West Nile Virus) by NAT or per current panel - must be negative for HIV and active hepatitis B
* Not pregnant - females of childbearing potential must have a negative pregnancy test within 7 days of apheresis
* Able and willing to undergo apheresis
* Voluntary written consent (using assent form if donor < 18 years of age)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of any grade 4 or greater suspected adverse reaction | 24 hours post infusion
Occurrence of Grade III or IV acute graft-versus-host disease (aGVHD) | 28 days post infusion

SECONDARY OUTCOMES:
Occurrence of treatment related mortality (TRM) | 2 months post infusion
Occurrence of disease response | 28 days post infusion
Number of patients alive without progression | 1 year post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cichocki F, Zhang B, Wu CY, Chiu E, Day A, O'Connor RS, Yackoubov D, Simantov R, McKenna DH, Cao Q, Defor TE, Janakiram M, Wangen R, Cayci Z, Snyder N, Kumar A, Grzywacz B, Hwang J, Geffen Y, Miller JS, Maakaron J, Bachanova V. Nicotinamide enhances natural killer cell function and yields remissions in patients with non-Hodgkin lymphoma. Sci Transl Med. 2023 Jul 19;15(705):eade3341. doi: 10.1126/scitranslmed.ade3341. Epub 2023 Jul 19. PMID 37467318